CLINICAL TRIAL: NCT05078814
Title: The Prevalence Survey of ALDH Gene Family in Patients With Peripheral Arterial Occlusive Disease or Acute Coronary Syndrome
Status: Recruiting | Type: Observational
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, Wei-Ting Chang, Doctor of Medicine, Chimei Medical Center
Other Study IDs: CMMC10705-003
Record Dates: First submitted 2021-09-06; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Artery Occlusive Disease; Acute Coronary Syndrome
Keywords: Peripheral Artery Occlusive Disease or Acute Coronary Syndrome
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational research — Observational research

SUMMARY:
Aldehyde dehydrogenase 2 (ALDH2) is an important enzyme protecting human from the accumulation of aldehyde, the main metabolites of alcohol. The deficiency of ALDH2 gene results in flush and hang over post drinking and most importantly it has been found associated with the incidence of cancer and post myocardial infarction (MI) heart failure. In the previous studies, ALDH2 decreased the ischemic territory post infarction and using a large scaled interaction of genetic variants and ALDH2 as an instrument, the threats of alcohol consumption on Asians' cardiovascular health was underscored. Furthermore, in a meta-analysis reviewing 12 case-control studies also indicated an increase of 48% risks in patients with ALDH2 deficiency. Notably, the genetic deficiency is most prevalent in Asians. In Taiwan one of every two individuals may be the victim and the high prevalence is counted as the top of the world. However, a large scaled prospective study focusing on the prevalence of ALDH2 deficiency in patients with peripheral artery occlusive disease (PAOD) or acute coronary syndrome （ACS）remains lacking.

ELIGIBILITY:
Inclusion Criteria:

1. Age≧20 y/o
2. Using ankle-brachial index (ABI)< 0.9, angiography, vascular duplex, CAT scan or cardiologists'impression to confirm the diagnosis of PAOD
3. Clinical presentation of claudication
4. diagnosis of ACS

Exclusion Criteria:

* If the patient refuses to be included in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed as peripheral arterial obstruction or acute coronary syndrome.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of MALE(major adverse limb events) in peripheral arterial disease and acute coronary disease. | 2 years

SECONDARY OUTCOMES:
The incidence of MACCE(major adverse cardiac and cerebrovascular events) in peripheral arterial disease and acute coronary disease. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Wei-Ting Chang, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No